CLINICAL TRIAL: NCT06841458
Title: Instrumental, Single-Blind, Placebo-Controlled Study Evaluating the Efficacy of a Dietary Supplement on Hair Growth Over 6 Months in 45 Volunteers
Brief Title: Six-Month Single-Blind, Placebo-Controlled Study of a Dietary Supplement Supplement on Hair Growth in 45 Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Industrial Farmacéutica Cantabria, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P24113a
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Androgenetic Alopecia
Keywords: MAGA; Androgenetic Alopecia; Natural supplement; Saw Palmetto; Cucurbita Pepo; Alopecia
MeSH Terms: conditions — Alopecia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Comparator (Placebo Comparator): Participants in the Placebo Comparator group will receive a placebo capsule identical in appearance to the active treatment but containing inactive ingredients with no known effect on hair growth. The intervention consists of one oral capsule per day for six months, administered under the same conditions as the active group.
  Interventions: Other: Oral Supplement
- Active Comparator (Active Comparator): Participants in the Active Comparator group will receive a dietary supplement designed to manage androgenetic alopecia (AGA). The intervention consists of one oral capsule per day for six months, containing active ingredients such as Saw Palmetto, Pumpkin Seed Oil, Pygeum africanum, L-Cystine, Oleanolic Acid, and Horsetail Extract.
  Interventions: Other: Oral Supplement

INTERVENTIONS:
Other: Oral Supplement — Participants in the Active Comparator group will receive a dietary supplement designed to manage androgenetic alopecia (AGA). The intervention consists of one oral capsule per day for six months, containing active ingredients such as Saw Palmetto, Pumpkin Seed Oil, Pygeum africanum, L-Cystine, Oleanolic Acid, and Horsetail Extract.

SUMMARY:
This clinical study is designed to evaluate the efficacy and safety of a dietary supplement CL-P24113a for the management of androgenetic alopecia (AGA) in male subjects aged 18 to 45 years who suffer from alopecia with low hair density, classified as mild to moderate (Hamilton-Norwood stages II, III, and IV). The product is a formulation based on a blend of botanical ingredients and other well-established compounds, including Pumpkin Seed Oil (Curcubita pepo), Saw Palmetto Oil (Serenoa repens), L-Cystine, Prunus africana Bark Extract (Pygeum africanum), Horsetail Extract (Equisetum arvense), Olive Leaf Extract, among other excipients. These components have a well-documented history of safe use in both topical and oral applications with supporting safety information from international bodies such as EFSA. In this instrumental, single-blind, placebo-controlled study, 45 volunteers will be divided into two groups, with 30 subjects receiving the supplement and 15 subjects receiving a placebo. All participants will ingest one capsule per day, preferably in the morning with a glass of water, over a 6-month treatment period. Prior to study initiation, subjects must complete a 30-day washout period using a neutral shampoo and agree not to apply any other topical or oral hair treatments in the target area throughout the study. The study will evaluate efficacy through both instrumental and subjective assessments. Instrumental evaluations will be conducted at 3 and 6 months using the TrichoScan HD Professional 4.0 system to measure hair growth parameters such as total hair count, hair density per cm², proportion of hairs, terminal hair count and density, proportion of terminal hairs, as well as the percentages of anagen and telogen hairs. Additionally, measurements of hair thickness including hair mass per cm², median and mean hair thickness in micrometers, overall scalp hair density, and median hair length will be recorded. Subjective evaluations will be performed via questionnaires administered at 1.5, 3, 4.5, and 6 months to capture participants' perceptions regarding hair growth and hair loss. The study is overseen by Principal Investigator at Dermaclaim Lab S.L. Regulatory compliance will be ensured by obtaining written informed consent for both study participation and data protection, and all subjects will be thoroughly briefed on study requirements and potential risks. This study aims to provide robust clinical evidence on the effectiveness of the oral supplement in promoting hair growth and reducing hair loss in men affected by androgenetic alopecia, potentially offering a safe and well-tolerated alternative to existing hair loss therapies while ensuring continuous monitoring for any adverse events throughout the treatment period.

DETAILED DESCRIPTION:
Nutraceutical foods are those that provide health benefits beyond basic nutrition. These include naturally occurring foods such as fish and vegetables, as well as processed foods like wine, yogurt, and dairy products. These natural compounds or substances exert therapeutic effects on the body, with the term 'nutraceutical' originating from the combination of 'nutrition' and 'therapeutic'

The classification of nutraceuticals is diverse and extensive, encompassing isolated nutrients, herbal products, fruit-derived supplements, dietary supplements, genetically modified foods, and processed products such as cereals, soups, and beverages . This diversity has enabled nutraceuticals to be widely available in commercial products spanning the food, pharmaceutical, herbal, and agro-industrial sectors.

One area of particular interest in nutraceutical research is hair health. The product to study has been developed to manage acute hair loss and to strengthen hair and nails. Thanks to its composition, including L-Cystine, glutathione, vitamins B5 and B6, copper, and zinc, it helps maintain hair and nail health. A new formulation of the product has been designed specifically to improve androgenetic alopecia (AGA) by incorporating natural ingredients that functionally inhibit the 5α-reductase enzyme.

Androgenetic alopecia (AGA) is one of the most common forms of hair loss in both men and women . It is characterized by the miniaturization of hair follicles due to the action of dihydrotestosterone (DHT) on androgen receptors. DHT is derived from testosterone via the 5α-reductase enzyme, which exists in three isoenzymes (types I, II, and III). Type II is most relevant to AGA as it is predominantly found in hair follicles. Many pharmacological interventions for AGA focus on inhibiting DHT's action on the hair follicle. Additionally, various molecules and vitamins are involved in the pathogenesis of AGA and in maintaining the proper cycle and structure of the hair follicle. The rationale for this study is based on the premise that the combination of different natural active ingredients inhibiting the 5α-reductase enzyme can work synergistically to improve signs associated with androgenetic alopecia. Serenoa Repens (Saw Palmetto) Cucurbita Pepo (Pumpkin Seed Oil) Pygeum Africanum Extract L-Cystine Oleanolic Acid Horsetail Extract (Equisetum arvense)

This observational study will evaluate the effects of the product in 30 volunteers receiving the active supplement and 15 receiving a placebo. The primary objective is to determine the supplement's effectiveness on hair health, growth, and hair loss over six months through instrumental (TrichoScan HD Professional 4.0) and subjective (questionnaires) evaluations. The study population consists of 45 male volunteers aged 18 to 45 years with hair growth and loss issues. The study will be conducted in compliance with regulatory guidelines, with careful monitoring of any potential adverse effects to ensure the safety and efficacy of the supplement.

Given that the key active ingredients in the product of study have established safety profiles and are widely used in commercial products, no significant adverse effects are anticipated. However, continuous monitoring will be conducted throughout the study to ensure participant safety and product efficacy. Volunteers will be compensated accordingly for their participation, and the study will be conducted under strict ethical and legal guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Written consent for LOPD compliance.
* Written informed consent for study DC.506.36.117.
* Gender: Male.
* Age: Between 18 and 45 years.
* Diagnosis of alopecia with low hair density, classified as mild to moderate (stages II, III, and IV on the Hamilton-Norwood scale).

Willingness to have a 1-2 cm² area shaved throughout the study period.

* Last participation in a clinical study on hair health must have ended at least six months before the start of this study.
* 30-day washout period without specific hair treatments (using a neutral shampoo).
* No use of any other topical or oral hair treatments in the target area during the study period; if necessary, consultation with the principal investigator is required to evaluate continued study participation.

Exclusion Criteria:

* Individuals with gastrointestinal diseases (e.g., diabetes, gastritis, Crohn's disease, celiac disease, ulcers, intolerances, etc.).
* Individuals with other physiological disorders (e.g., diabetes, hypertension, dyslipidemia) and/or gallstones.
* Individuals undergoing medical treatment in the weeks prior to the study that may interfere with study assessments (as determined by the investigator), particularly those who are currently taking or have taken 5α-reductase inhibitors (Finasteride, Dutasteride, Minoxidil, etc.) within the last three months.

Individuals who have undergone hair restoration treatments at any point in their lives, including hair transplants, mesotherapy, or platelet-rich plasma (PRP) therapy.

* Individuals following an atypical diet or planning to change their dietary routine during the study period.
* Individuals enrolled in another clinical study with similar characteristics (as determined by the investigator) during the study period.
* Individuals who are unable to fully understand the informed consent document or adhere to the study protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Evaluation of Hair Health Benefits After Six Months of Treatment | From enrollment to 3 months and 6 months
  Hair Growth Assessment Using Phototrichogram Analysis
  Description: Evaluation of hair growth parameters using the TrichoScan HD Professional 4.0 system. The analysis will be performed 48 hours after shaving a 1 cm² region of interest (ROI). The following parameters will be measured:
  1-Total Hair Count: number of hairs in 1 cm². Unit= number of hairs
Total Terminal Count | From enrollment to 3 months and 6 months
  Total Terminal Count: # terminal hairs. Unit= number of hairs
Hair Density | From enrollment to 3 months and 6 months
  Hair Density: hairs/cm². Unit=hairs/cm²
Terminal Hair Density | From enrollment to 3 months and 6 months
  Terminal Hair Density: terminal hairs/cm². Unit=hairs/cm²
Terminal Hair Proportion | From enrollment to 3 months and 6 months
  Terminal Hair Proportion: % of terminal hairs. Unit=%
Anagel and Telogen | From enrollment to 3 months and 6 months
  Anagen %: anagen. Unit=% Telogen %: telogen. Unit=%
Hair Mass | From enrollment to 3 months and 6 months
  Hair Mass: mm/cm². Unit=mm/cm²
Median and Mean Hair Thickness | From enrollment to 3 months and 6 months
  Median Hair Thickness: μm. Unit=μm Mean Hair Thickness: μm. Unit=μm
Hair length | From enrollment to 3 months and 6 months
  Hair Length: average length. Unit=mm or cm

SECONDARY OUTCOMES:
Subjective evaluation questionnaire | From enrollment to 3 months and 6 months
  Consumer perception of the dietary supplement will be analyzed, including its organoleptic properties, efficacy and functionality, and consumption characteristics.
  The scale used in this subjective self-assessment questionnaire is a 4-point Likert scale with the following values: 1 = Strongly disagree, 2 = Disagree, 3 = Agree, and 4 = Strongly agree. A favorable response is defined as selecting either 3 (Agree) or 4 (Strongly Agree). This scale measures the participant's subjective experience regarding the treatment. A higher score indicates a more positive perception of the treatment outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - DermaClaim, Valencia, Valencia
  - DermaClaim, Valencia

IPD SHARING:
Plan to Share IPD: No